CLINICAL TRIAL: NCT04930978
Title: Effect of SARS-CoV-2 Disease on Immune Responses, Disease Severity and Treatment Outcomes in Pulmonary Tuberculosis
Acronym: COVID-19-TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tuberculosis Research Centre, India (Other Government)
Responsible Party: Principal Investigator, Dr. S. Subash Babu, Scientific Director, Tuberculosis Research Centre, India
Other Study IDs: 2020 041
Record Dates: First submitted 2021-06-12; First posted 2021-06-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Respiratory Infection; Pulmonary Tuberculoses
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A portion of the samples (serum, cells) of each subject will be stored for future research, after obtaining informed consent from the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TB patients with SARS-CoV-2 PCR+: 50 TB patients with SARS-CoV-2 PCR+ will be recruited in group 1
- TB patients with SARS-CoV-2 Ab+: 100 TB patients with SARS-CoV-2 Ab+ will be recruited in group 2
- TB patients negative for SARS-CoV-2 PCR and Ab: 100 TB patients with SARS-CoV-2 PCR and Ab negative will be recruited in group 3

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the causative agent of the Coronavirus disease (COVID-19). Tuberculosis (TB) is the foremost cause of infectious deaths globally. In 2025, an additional 1.4 million TB deaths could occur as direct consequence of the COVID-19 pandemic. It is postulated that individuals with latent or active TB are more susceptible to SARS-CoV-2 disease and that COVID-19 disease rate is high in patients with active TB, although the evidence is still scarce. TB and SARS-CoV-2 are both infectious diseases which primarily attack the alveolar region of the lungs and share common symptoms. SARS-CoV-2 disease can induce innate and adaptive immunity, but uncontrolled inflammatory innate immunity and impaired adaptive immune responses may be associated with severe tissue damage, both locally and systemically. People with coinfection (COVID-19 and TB disease) might potentially have impaired protective immune responses and treatment outcomes, specifically as far as anti-tuberculosis treatment is concerned. However, very little is known about the immunological underpinnings in this interface between TB and COVID-19 on the effect of SARS-CoV-2 disease on disease severity, response to treatment and treatment outcomes in pulmonary tuberculosis. Investigators hypothesize that altered immunity due to prior or present asymptomatic disease with SARS-CoV-2 virus can lead to altered immune responses and systems biology, increased severity and altered treatment outcomes in TB disease.

The main objective of the study would be to evaluate the baseline differences in immune cells populations immune cell responses at baseline and at the time of treatment (2nd month) and end of treatment. Further, Investigators would be evaluating the changes in proteomic profiles in a subset of these individuals. In addition, immunological assays examining differences in T cell populations, measuring levels of various cytokines and by immunophenotyping as well as other immune parameters related to innate and adaptive responses will be performed to enhance the understanding of the immunological cross-talk between active TB patients with or without SARS-CoV-2. The secondary objective would be to study the clinical features, disease severity, mycobacterial burden and treatment outcomes in a cohort of SARS-CoV-2 infected (asymptomatic PCR or Antibody+) and non-infected patients with active pulmonary TB.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is a new respiratory infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which belongs to the family coronaviridae with wide spreading in humans and animals. This virus is enveloped and contains positive-sense, single-stranded RNA with approximately 31 kb of genome size and so far, is considered as the largest known RNA viruses. The COVID-19 infected individuals exhibit low to modest symptoms (cough, fever, and respiratory distress) and transmitted mainly by respiratory droplets. However, around 15% of infected individuals proceed to severe pneumonia and approximately 5% of them progress to acute respiratory distress syndrome (ARDS), septic shock and/or multiple organ failure. Transmission of SARS-CoV-2 occurs through the means of coughing and sneezing, touching the mouth, nose, eyes, close personal contact and touching a virus-contaminated object. SARS-CoV-2 disease can induce both the arms of innate and adaptive immunity, but uncontrolled inflammatory innate immunity and weakened adaptive immune responses might be associated with destructive tissue damage, both locally and systemically. Patients with severe COVID-19 exhibited decrease of lymphocytes, and the elevation of IL-6, IL-10 and C-reactive protein. The SARS-CoV-2 is a global pandemic threat. Currently, as on August 5, the total number of COVID-19 cases is approximately 18,354,342 with 696147 deaths were reported worldwide and 216 countries are affected. In India, approximately 1,908,254 individuals were infected and 39795 deaths occurred due to COVID-19. SARS-CoV-2 disease is often associated with unconstrained immune response, caused by the hyperactivation of monocytes, macrophages and elevated neutrophils. Both, humoral (production of IgG, IgM, neutralising antibodies and reduced memory B cells) and cell mediated (CD4+, CD8+ and cytotoxic markers) immunity is required for defense against COVID-19. In addition, the activation of Th1 / Th17 cells might induce the exacerbation of the inflammatory response.

Tuberculosis (TB) is one of the most important infectious diseases around the world. Tuberculosis (TB), although largely a curable disease, still remains a major cause of morbidity and mortality worldwide. According to the Global Tuberculosis Report 2019, there are an estimated 10 million incident cases of tuberculosis and killed 1.2 million in 2018 globally. India accounts for 27% of all estimated incident cases worldwide. M. tuberculosis (M.tb) infection could result in the activation of innate (monocytes, macrophages, dendritic cells, neutrophils, mast cells) and adaptive (CD4+ and CD8+ T cells, cytotoxic markers) immune response which are necessary for protection. Protective immunity against M. tuberculosis is not completely understood but depends on a wide range of innate and adaptive immune mechanisms. T cell-mediated immune responses are important in the host control of M. tuberculosis infection. The ability of CD4+ T cells to produce gamma interferon, which activates phagocytes to contain the intracellular pathogen, is central in protection. Indeed, T helper 1 (Th1) cells and the gamma IFN that they produce are crucial for protection against disease. This is evident from the increased risk of tuberculosis in individuals with deficiencies in their IFNγ and interleukin 12 (IL 12; which promotes Th1 cell differentiation) signalling pathways. Many other CD4+ T cell subsets, in addition to gamma IFN producing Th1 cells, may also have a role; for example, IL 17-producing CD4+ T cells were shown to mediate the recruitment of protective Th1 cells to the lung upon M. tuberculosis challenge. Furthermore, increased frequencies of regulatory CD4+ T regulatory (Treg) cells during active disease may ensure that the Th1 cell response is not excessive, and this would help minimize lung damage in tuberculosis. The CD8+ T cell response to M. tuberculosis is normally of a lower magnitude than the CD4+ T cell response; however, CD8+ T cells may modulate phago¬cyte activity or produce molecules such as granulysin that may be directly cytotoxic to the mycobacteria. Similarly, other cytokines, in addition to gamma IFN, may also be crucial; for example, Tumour necrosis factor-alpha is important for establishing the granuloma, which is a well-organized collection of innate and adaptive cells that forms to contain the pathogen. Development of TB disease results from interactions among the environment, the host, and the pathogen, and known risk factors include HIV coinfection, immunodeficiency, diabetes mellitus, overcrowding, malnutrition, and general poverty.

The link between TB and COVID-19 is likely to be bi-directional. The temporary immunosuppression induced by tuberculosis may increase the susceptibility of patients to COVID-19, and COVID may, in turn, also increase susceptibility to TB. In 2025, an additional 1.4 million TB deaths could be occurred as direct consequence of the COVID-19 pandemic. The COVID-19 disease rate was high in patients with active TB. TB and SARS-CoV-2 are both infectious diseases which primarily attack the alveolar region of the lungs and share common symptom patterns. Both CD4 and CD8 counts were severely reduced, and the surviving T cells appeared to demonstrate "functional exhaustion". This T cell depletion and dysfunction may exacerbate active TB. Published studies have reported that patients with TB and other viral infections impede the host immune responses like induction of type I interferons by influenza infection, lower mean of CD4+ and CD8+ T cells and increased viral elimination in sputum, stool and suppression of cellular immunity. Recent studies have reported that cytokines seem to play an important role in COVID-19 and TB, and their plasma levels associated with disease severity. It is predicted that people with coinfection have impaired protective immune responses and treatment outcomes, specifically in terms of anti-tuberculosis treatment. Studies showed that SARS-CoV2 coexistent with TB resulted in a decreased absolute number of CD4+ and CD8+ T cells and reduced antibody levels following SARS-CoV-2 recovery. SARS-CoV-2 with TB patients exhibited prolonged viral elimination from stools and sputum in comparison without TB. Studies have demonstrated that SARS-CoV-2 disease stimulates increased cytokine secretion, like interleukin-1 , gamma interferon, tumour necrosis factor- alpha, interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-10 (IL-10), that ultimately leads to severe inflammation and their plasma levels were linked with disease severity. However, only limited information is available on the function of antigen-specific T cell-mediated immune response to COVID-19 specifically upon coinfection with tuberculosis, since both the disease primarily affects the lungs.

Limited studies have shown that influenza induces immune system hyperactivity and exacerbates pulmonary tuberculosis, leading to worsening of pulmonary function. Respiratory viral infections coexistent with TB delay the host immune responses and lead to more serious clinical outcomes. Coinfection most probably exacerbates inflammation through heightened secretion of cytokines and accelerates the development of severe acute respiratory syndrome and also worsen the TB disease and its outcome. Hence, Investigators propose that understanding mechanisms of immune regulation during SARS-CoV-2 disease may lead to the development of better therapeutic strategies and the results of our fundamental studies may inform future plans for clinical interventional studies. The main fundamental research component of this study might identify clinical parameters and treatment methods and to understand the immunological mechanism for the severity in coinfected SARS-CoV-2 and TB patients.

Hypothesis: Investigators hypothesize that altered immunity due to present or prior asymptomatic disease with SARS-CoV-2 virus could lead to altered immune responses and systems biology, increased severity and altered treatment outcomes in TB disease.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-65;
* Newly diagnosed smear or GeneXpert positive for TB with or without SARS-CoV-2 (present or prior asymptomatic) disease;
* Willing to provide written informed consent.

Exclusion Criteria:

* Any prior episode of TB disease;
* Treatment for current TB episode >1 week before enrollment;
* Drug resistance TB patients;
* Pregnancy or childbirth within last 6 months;
* Diabetes, HIV-seropositive and current use of immunosuppressive and steroid therapy Mild, Moderate and severe Covid-19 disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of SARS-CoV-2 via RT-PCR or antibody testing. Diagnosis of TB and classification of TB treatment outcomes are as per National Tuberculosis Elimination program definitions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with active TB | Day 1
  Effects of SARS-CoV-2 on TB severity, altered Immunological and systems biological Measured by smear or GeneXpert
Number of participants with COVID-19 infection | Day 1
  Measured by real-time qPCR (quantitative polymerase chain reaction) assay
Number of participants with SARS-CoV-2 antibodies | Day 1
  Measured by SARS-CoV-2 serology
Differences in immune responses between the groups | 2 years
  Measured by immunological assays

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Rajamanickam, PhD, Principal Investigator — National Institute for Research in Tuberculosis-International Centers for Excellence in Research
Locations (1):
- National Institute for Research in Tuberculosis, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No